CLINICAL TRIAL: NCT01579916
Title: A Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Safety of 3 New 6:2 Influenza Virus Reassortants in Adults
Brief Title: A Study to Evaluate the Safety of 3 New 6:2 Influenza Virus Reassortants in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CD-VA-FluMist-1114
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2013-12

CONDITIONS: Influenza
Keywords: Trivalent, Influenza, FluMist, Vaccine, Prevention
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trivalent Influenza Virus Vaccine (Experimental): Trivalent vaccine is supplied in intranasal sprayers containing a total volume of 0.5 mL of sucrose phosphate buffer, egg allantoic fluid and approximately 10^7 FFU (fluorescent focus units) of each of 3 cold-adapted, attenuated 6:2 reassortant influenza strains: A/H1N1 (A/California/7/2009), A/H3N2 (A/Victoria/361/2011), B (B Wisconsin/1/2010). A single dose of investigational product was administered on Day 1.
  Interventions: Biological: Trivalent Influenza Virus Vaccine
- Placebo (Placebo Comparator): Placebo is suppllied in intranasal sprayers containing 0.5 mL of sucrose-phosphate buffer. A single dose of investigational product was administered on Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Trivalent Influenza Virus Vaccine — Trivalent vaccine is supplied in intranasal sprayers containing a total volume of 0.5 mL of sucrose phosphate buffer, egg allantoic fluid and approximately 10^7 FFU (fluorescent focus units) of each of 3 cold-adapted, attenuated 6:2 reassortant influenza strains: A/H1N1 (A/California/7/2009), A/H3N2 (A/Victoria/361/2011), B (B Wisconsin/1/2010). A single dose of investigational product was administered on Day 1.
  Arms: Trivalent Influenza Virus Vaccine
Other: Placebo — Placebo is suppllied in intranasal sprayers containing 0.5 mL of sucrose-phosphate buffer. A single dose of investigational product was administered on Day 1.
  Arms: Placebo

SUMMARY:
This prospective annual release study was designed to assess the safety of a trivalent influenza virus vaccine using two new strains recommended for the 2012-2013 influenza season not previously contained in the trivalent intranasal FluMist vaccine.

Three hundred healthy adults will receive a single dose of vaccine or placebo and will be followed for 180 days after study vaccination.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, placebo-controlled release study will enroll approximately 300 healthy adults 18 to 49 years of age. Eligible subjects will be randomly assigned in a 4:1 fashion to receive a single dose of trivalent vaccine or placebo by intranasal spray. Randomization will be stratified by site.

This study will be conducted at 3 sites in the United States of America. Each subject will receive one dose of investigational product on Study Day 1. The duration of study participation for each subject is the time from study vaccination through 180 days after study vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 49 years at the time of investigational product administration
2. Written informed consent and any locally required authorization (ie, HIPAA in the USA) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
3. Females of childbearing potential who are sexually active with a nonsterilized male partner must use effective contraception for 30 days prior to study vaccination, and must agree to continue using such precautions for 60 days after study vaccination
4. Nonsterilized males who are sexually active with a female partner of child-bearing potential must use an effective method of contraception from prior to study vaccination amd must agree to continue using such precautions for at least 30 days after receipt study vaccination
5. Healthy by medical history and physical examination
6. Female subjects of child-bearing potential must also have a negative urine or blood pregnancy test at screening and, if screening and Day 1 do not occur on the same day, on the day of vaccination prior to randomization.
7. Subject available by telephone
8. Ability to understand and comply with the requirements of the protocol, as judged by the investigator
9. Ability to complete follow-up period of 180 days after dosing as required by the protocol

Exclusion Criteria:

1. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
2. Concurrent enrollment in another clinical study up to 180 days after receipt of investigational product (Day 181)
3. Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals
4. History of hypersensitivity to any component of the vaccine, including egg or egg protein or serious, life threatening, or severe reactions to previous influenza vaccinations
5. History of hypersensitivity to gentamicin
6. Any condition for which the inactivated influenza vaccine is indicated, including chronic disorders of the pulmonary or cardiovascular systems (eg, asthma), chronic metabolic diseases (eg, diabetes mellitus), renal dysfunction, or hemoglobinopathies that required regular medical follow-up or hospitalization during the preceding year
7. Acute febrile (> 100.0°F oral or equivalent) and/or clinically significant respiratory illness (eg, cough or sore throat) within 14 days prior to randomization
8. Any known immunosuppressive condition or immune deficiency disease, including human immunodeficiency virus infection, or ongoing immunosuppressive therapy
9. History of Guillain-Barré syndrome
10. A household contact who is severely immunocompromised (eg, hematopoietic stem cell transplant recipient, during those periods in which the immunocompromised individual requires care in a protective environment); additionally, subject should avoid close contact with severely immunocompromised individuals for at least 21 days after study vaccination
11. Receipt of any investigational agent within 30 days prior to randomization, or expected receipt through 30 days after study vaccination (use of licensed agents for indications not listed in the package insert is permitted)
12. Receipt of any non-study vaccine within 30 days prior to randomization, or expected receipt through 30 days after study vaccination
13. Expected receipt of antipyretic or analgesic medication on a daily or every other day basis from randomization through 14 days after study vaccination
14. Administration of intranasal medications within 14 days prior to randomization, or expected receipt through 14 days after study vaccination
15. Receipt of influenza antiviral therapy or antiviral agents within 48 hours prior to study vaccination or expected receipt of influenza antiviral therapy or antiviral agents through 14 days after study vaccination
16. Known or suspected mitochondrial encephalomyopathy
17. Nursing mother

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 303 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raburn Mallory, MD, Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Research Site, Miami, Florida
  - Research Site, Stockbridge, Georgia
  - Research Site, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 303 participants participated in the study from 21May2012 (date of first written informed consent) through 30Nov2012 (date of last participant visit).
Pre-assignment Details: Eligible participants were randomly assigned in a 4:1 fashion to receive a single dose of trivalent vaccine or placebo by intranasal spray. Randomization was stratified by site.
Groups:
- Placebo: Placebo is supplied in intranasal sprayers containing 0.5 mL of sucrose-phosphate buffer. A single dose of investigational product was administered on Day 1.
Period: Overall Study
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Started | 242 | 61
Completed | 234 | 59
Not Completed | 8 | 2
Not completed — Lost to Follow-up | 6 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo | TOTAL
Number analyzed (Participants) | 242 | 61 | 303
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.7 (9.1) | 32.0 (8.8) | 32.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 29 | 165
  Male | 106 | 32 | 138

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Fever Within 7 Days Post Vaccination
Description: A comparison of the rate of fever, defined as oral temperature greater than or equal to 101 degrees Fahrenheit, reported during the 7 days post administration of investigational product between the trivalent influenza virus vaccine and placebo groups.
Time Frame: Study Days 1 - 8
Population: All participants who received a single dose of investigational product (trivalent influenza vaccine = 241; placebo = 60).
Measure: Number; unit: Percentage of Participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 241 | 60
Percentage of Participants | 0.0 | 1.7
Statistical Analysis 1: Comparison: Trivalent Influenza Virus Vaccine vs Placebo; Comparison of the rate of fever between the 2 treatment groups was based on the upper limit of the two-sided 95% exact confidence intervals (CIs) for the rate increase (trivalent influenza virus vaccine minus placebo) evaluated against the prespecified equivalence criterion of 5 percentage points; Test type: Non-Inferiority or Equivalence — H0 (null): Rate difference greater than or equal to 5 percentage points. This corresponds to a null hypothesis of: HA (alternative): rate difference < 5 percentage points; Score statistic; Rate difference = -1.7, 95% CI 2-sided [-8.9 to 0.6]

2. Secondary Outcome: Percentage of Participants Reporting Other Solicited Symptoms Within 7 Days Post Vaccination
Description: Solicited symptoms were events that were considered likely to occur post dosing. Solicited symptoms for this study are listed below.
Time Frame: Study Days 1- 8
Population: All participants who received a single dose of investigational product (trivalent influenza virus vaccine = 241; placebo = 60)
Measure: Number; unit: Percentage of Participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 241 | 60
Percentage of Participants
  Any symptom | 38.6 | 20.0
  Fever > 100 degrees Fahrenheit | 0.8 | 1.7
  Fever >/= 101 degrees Fahrenheit | 0.0 | 1.7
  Fever > 102 degrees Fahrenheit | 0.0 | 0.0
  Fever > 103 degrees Fahrenheit | 0.0 | 0.0
  Runny nose | 18.3 | 8.3
  Sore throat | 14.1 | 5.0
  Cough | 4.1 | 1.7
  Vomiting | 0.4 | 0.0
  Muscle aches | 5.0 | 3.3
  Chills | 1.2 | 3.3
  Decreased activity (tiredness) | 8.7 | 6.7
  Headache | 15.8 | 10.0

3. Secondary Outcome: Percentage of Participants Reporting Any Adverse Event (AE) Within 7 Days Post Vaccination
Description: Percentage of participants reporting at least one AE between Days 1 and 8. Investigational product was administered on Day 1.
Time Frame: Study Days 1 - 8
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 241 | 60
Percentage of participants | 7.5 | 6.7

4. Secondary Outcome: Percentage of Participants Reporting Other Solicited Symptoms Within 14 Days Post Vaccination
Description: as for outcome 2
Time Frame: Study Days 1 - 15
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 241 | 60
Percentage of participants
  Perecentage of participants reporting any symptom | 41.5 | 25.0
  Fever > 100 degrees Fahrenheit | 1.2 | 1.7
  Fever >/= 101 degrees Fahrenheit | 0.4 | 1.7
  Fever > 102 degrees Fahrenheit | 0.0 | 0.0
  Fever > 103 degrees Fahrenheit | 0.0 | 0.0
  Runny nose | 19.1 | 13.3
  Sore throat | 14.9 | 5.0
  Cough | 5.4 | 3.3
  Vomiting | 0.4 | 0.0
  Muscle aches | 5.8 | 3.3
  Chills | 1.2 | 3.3
  Decreased activity (tiredness) | 8.7 | 8.3
  Headache | 17.4 | 11.7

5. Secondary Outcome: Percentage of Participants Reporting Any Adverse Event (AE) Within 14 Days Post Vaccination
Description: Percentage of participants reporting at least one AE between Days 1 and 15. Investigational product was administered on Day 1.
Time Frame: Study Days 1 - 15
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 241 | 60
Percentage of participants | 7.9 | 6.7

6. Secondary Outcome: Percentage of Participants Reporting Any Serious Adverse Event (SAE) Within 28 Days Post Vaccination
Description: Percentage of participants reporting at least one SAE between Days 1 and 29. Investigational product was administered on Day 1.
Time Frame: Study Days 1 - 29
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 241 | 60
Percentage of participants | 0.0 | 0.0

7. Secondary Outcome: Percentage of Participants Reporting Any Serious Adverse Event (SAE) Within 180 Days Post Vaccination
Description: Percentage of participants reporting at least one SAE between Days 1 and 181. Investigational product was administered on Day 1.
Time Frame: Study Days 1 - 181
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 241 | 60
Percentage of participants | 0.4 | 1.7

8. Secondary Outcome: Percentage of Participants Reporting Any New Onset Chronic Diseases (NOCDs) Within 28 Days Post Vaccination
Description: An NOCD was a newly diagnosed medical condition of a chronic, ongoing nature and assessed by the investigator as medically significant. Such events were assessed between Day 1 and Day 29. Investigational product was administered on Day 1.
Time Frame: Study Days 1 - 29
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 241 | 60
Percentage of participants | 0.0 | 0.0

9. Secondary Outcome: Percentage of Participants Reporting Any New Onset Chronic Diseases (NOCDs) Within 180 Days Post Vaccination
Description: An NOCD was a newly diagnosed medical condition of a chronic, ongoing nature and assessed by the investigator as medically significant. Such events were assessed between Day 1 and Day 181. Investigational product was administered on Day 1.
Time Frame: Study Days 1 - 181
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 241 | 60
Percentage of participants | 0.4 | 0.0

10. Secondary Outcome: Percentage of Participants Who Used Antipyretic or Analgesic Agents Within 7 Days Post Vaccination
Description: Percentage of participants who used an antipyretic or analgesic agent between Days 1 and 8. Investigational product administration occurred on Day 1.
Time Frame: Study Days 1 - 8
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 241 | 60
Percentage of Participants | 2.1 | 3.3

11. Secondary Outcome: Percentage of Participants Who Used Antipyretic or Analgesic Agents Within 14 Days Post Vaccination
Description: Percentage of participants who used an antipyretic or analgesic agent between Days 1 and 15. Investigational product administration occurred on Day 1.
Time Frame: Study Days 1 - 15
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 241 | 60
Percentage of Participants | 2.1 | 3.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of investigational product administration through Day 15. Serious adverse events were collected from the time of study drug administration through Day 181.
Arm/Group | Trivalent Influenza Virus Vaccine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/241 | 1/60
Other Adverse Events (participants affected / at risk) | 19/241 | 4/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trivalent Influenza Virus Vaccine (N=241) | Placebo (N=60)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trivalent Influenza Virus Vaccine (N=241) | Placebo (N=60)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.